CLINICAL TRIAL: NCT01160289
Title: A Study of LY900010 (LY2452473 + Tadalafil) in the Treatment of Men With Erectile Dysfunction
Brief Title: A Study of LY900010 in Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11888; I4K-MC-GPEC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — LY2452473; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 milligram (mg) LY2452473 + 5 mg tadalafil (Experimental)
  Interventions: Drug: LY2452473; Drug: tadalafil; Drug: placebo (tadalafil)
- 5 mg LY2452473 + 5 mg tadalafil (Experimental)
  Interventions: Drug: LY2452473; Drug: tadalafil; Drug: placebo (tadalafil)
- 5 mg LY2452473 + placebo (Experimental)
  Interventions: Drug: LY2452473; Drug: placebo (tadalafil)
- 10 mg tadalafil + placebo (Active Comparator)
  Interventions: Drug: tadalafil; Drug: placebo (tadalafil); Drug: placebo (LY2452473)
- 5 mg tadalafil + placebo (Active Comparator)
  Interventions: Drug: tadalafil; Drug: placebo (tadalafil); Drug: placebo (LY2452473)

INTERVENTIONS:
Drug: LY2452473 — Administered orally, once daily for 12 weeks
  Arms: 1 milligram (mg) LY2452473 + 5 mg tadalafil; 5 mg LY2452473 + 5 mg tadalafil; 5 mg LY2452473 + placebo
Drug: tadalafil — Administered orally, once daily for 12 weeks
  Arms: 1 milligram (mg) LY2452473 + 5 mg tadalafil; 10 mg tadalafil + placebo; 5 mg LY2452473 + 5 mg tadalafil; 5 mg tadalafil + placebo
Drug: placebo (tadalafil) — Administered orally, once daily for 12 weeks
Drug: placebo (LY2452473) — Administered orally, once daily for 12 weeks
  Arms: 10 mg tadalafil + placebo; 5 mg tadalafil + placebo

SUMMARY:
The primary purpose of the study is to compare the efficacy of LY2452473 + tadalafil to tadalafil alone in improving the erectile function (EF) of men with erectile dysfunction (ED) who incompletely respond to tadalafil alone.

ELIGIBILITY:
Inclusion Criteria include:

* Ambulatory men
* History of erectile dysfunction of at least 3 months duration
* History of incomplete response to any phosphodiesterase type 5 inhibitor (PDE5i) at the maximum tolerated dose within the label
* Anticipate having the same female sexual partner throughout the duration of the study
* Are willing and able to make at least 4 sexual intercourse attempts with the female sexual partner during each 4-week segment of the study
* Agree to use birth control during the study and for 60 days after the study, unless the female partner is postmenopausal
* Agree not to use any other erectile dysfunction treatment, including herbal treatment, during the study and for 96 hours after the last dose of study drug
* Screening laboratory tests within normal limits except for testosterone
* Without a language barrier, are reliable and willing to follow study procedures
* Prostate-specific antigen (PSA) less than 10 nanograms per milliliter (ng/ml). Men with PSA greater than 4 and less than 10 ng/ml must have documentation of a negative histological biopsy of carcinoma of prostate within 12 months prior to screening

Exclusion Criteria include:

* History of penile implant
* History of no response to injection therapy for erectile dysfunction
* History of radical prostatectomy or other pelvic surgery with subsequent failure to achieve any erection
* Exhibit the presence of clinically significant penile deformity in the opinion of the investigator
* History of prior sexual legal convictions
* Bilateral hip replacements
* History of cancer within the previous 5 years, except for excised superficial lesions such as basal cell carcinoma and squamous cell carcinoma of the skin
* Chronic stable angina currently treated with long-acting nitrates
* Chronic stable angina requiring treatment with short-acting nitrates within 90 days prior to screening
* Angina occurring during sexual intercourse in the 6 months prior to screening
* Unstable angina within 6 months prior to screening
* Myocardial infarction or coronary artery bypass graft surgery within 90 days prior to screening
* Angioplasty or stent placement within 90 days prior to screening
* Congestive heart failure within 6 months prior to screening
* History of sudden cardiac arrest
* Supraventricular arrhythmia with an uncontrolled ventricular response at rest, or any history of spontaneous or induced sustained ventricular tachycardia, or use an automatic internal cardioverter-defibrillator
* An abnormality in the 12-lead electrocardiogram (ECG) that in the opinion of the investigator places the subject in an unacceptable risk for study participation
* Systolic blood pressure greater than 170 or less than 90 millimeters of mercury (mm Hg) or diastolic blood pressure greater than 100 or less than 50 mm Hg at screening
* Hepatic, renal, human immunodeficiency virus (HIV), or clinically significant active neuropsychiatric disease
* History of central nervous system injuries (including stroke or spinal cord injury) within 6 months prior to screening
* Alcohol intake of 5 units or greater per day (1 unit = 12 ounces beer, 5 ounces wine, or 1.5 ounces of 80-proof distilled spirits)
* Receiving treatment with antiandrogens or 5-alpha reductase inhibitor
* Anabolic steroids, calcitonin, oral bisphosphonates, Vitamin D greater than 50,000 international units per week (IU/week), dehydroepiandrosterone (DHEA), steroidal supplements, nutritional products intended to have weight reduction or performance enhancing effects, herbal supplements within 7 days prior to screening
* Currently treated with a potent cytochrome P450 (CYP) 3A4 inhibitor, such as systemic ketoconazole or ritonavir, or a CYP3A4 inducer such as rifampicin

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (36):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendora, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vacaville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Englewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Celebration, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coeur d'Alene, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cary, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmond, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had 2 periods. Period 1: a screening, a 4-week washout, and a 4-week lead-in period prior to randomization. Period 2: a 12-week treatment and a 4-week follow-up period, post-randomization.
Groups:
- All Screened Subjects: After screening but prior to randomization, subjects completed a 4-week washout and a 4-week tadalafil [5-milligram (mg) tablet, administered orally, once daily] lead-in period.
- 1 mg LY2452473 and 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 1-mg capsule
  * tadalafil 5-mg tablet
  * placebo 10-mg tablet (matching tadalafil)
- 5 mg LY2452473 and 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 5-mg capsule
  * tadalafil 5-mg tablet
  * placebo 10-mg tablet (matching tadalafil)
- 5 mg LY2452473: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 5-mg capsule
  * placebo 5-mg tablet (matching tadalafil)
  * placebo 10-mg tablet (matching tadalafil)
- 10 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * tadalafil 10-mg tablet
  * placebo 5-mg capsule (matching LY2452473)
  * placebo 5-mg tablet (matching tadalafil)
- 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * tadalafil 5-mg tablet
  * placebo 5-mg capsule (matching LY2452473)
  * placebo 10-mg tablet (matching tadalafil)
Period: Screening, Washout, and Lead-In Period
Arm/Group | All Screened Subjects | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Started | 894 | 0 | 0 | 0 | 0 | 0
Completed | 410 | 0 | 0 | 0 | 0 | 0
Not Completed | 484 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 308 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 26 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization Criteria Not Met | 67 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 64 | 0 | 0 | 0 | 0 | 0
Period: Post-Randomization Period
Arm/Group | All Screened Subjects | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Started | 0 | 85 | 97 | 52 | 89 | 87
Received at Least 1 Dose of Study Drug | 0 | 85 | 97 | 52 | 89 | 87
Completed | 0 | 65 | 73 | 31 | 80 | 73
Not Completed | 0 | 20 | 24 | 21 | 9 | 14
Not completed — Adverse Event | 0 | 4 | 4 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 5 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 2 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 5 | 13 | 8 | 5 | 7
Not completed — Entry Criteria Not Met | 0 | 2 | 2 | 2 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 1 mg LY2452473 and 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 1-mg capsule
  * tadalafil 5-mg tablet
  * placebo 10-mg tablet (matching tadalafil)
  Prior to randomization, participants successfully completed a 4-week washout and a 4-week tadalafil (5-mg tablet, daily) lead-in period.
- 5 mg LY2452473 and 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 5-mg capsule
  * tadalafil 5-mg tablet
  * placebo 10-mg tablet (matching tadalafil)
  Prior to randomization, participants successfully completed a 4-week washout period and a 4-week tadalafil (5-mg tablet, daily) lead-in period.
- 5 mg LY2452473: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * LY2452473 5-mg capsule
  * placebo 5-mg tablet (matching tadalafil)
  * placebo 10-mg tablet (matching tadalafil)
  Prior to randomization, participants successfully completed a 4-week washout period and a 4-week tadalafil (5-mg tablet, daily) lead-in period.
- 10 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * tadalafil 10-mg tablet
  * placebo 5-mg capsule (matching LY2452473)
  * placebo 5-mg tablet (matching tadalafil)
  Prior to randomization, participants successfully completed a 4-week washout period and a 4-week tadalafil (5-mg tablet, daily) lead-in period.
- 5 mg Tadalafil: The following study drugs, administered orally, once daily for 12 weeks post-randomization:
  * tadalafil 5-mg tablet
  * placebo 5-mg capsule (matching LY2452473)
  * placebo 10-mg tablet (matching tadalafil)
  Prior to randomization, participants successfully completed a 4-week washout period and a 4-week tadalafil (5-mg tablet, daily) lead-in period.
- Total: Total of all reporting groups
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil | Total
Number analyzed (Participants) | 85 | 97 | 52 | 89 | 87 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.57) | 60.7 (6.57) | 58.7 (6.53) | 59.4 (6.54) | 60.5 (6.68) | 59.9 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 85 | 97 | 52 | 89 | 87 | 410
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 3 | 13 | 10 | 48
  Not Hispanic or Latino | 76 | 84 | 49 | 76 | 77 | 362
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 2 | 0 | 5
  Asian | 2 | 2 | 0 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 17 | 7 | 13 | 8 | 59
  White | 68 | 76 | 45 | 72 | 78 | 339
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 97 | 52 | 89 | 87 | 410

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF) Erectile Function (EF) Domain Score
Description: The IIEF EF domain score was the sum of Questions (Q) 1 to Q5 and Q15 of the IIEF self-reported questionnaire. Q1 to Q5 were rated 0 (low/no EF) to 5 (high EF) and Q15 was rated 1 (no/low confidence) to 5 (high confidence). IIEF EF domain scores ranged from 1 to 30. Higher scores denoted better EF.
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug [intention-to-treat (ITT) population] and had non-missing IIEF EF domain scores at baseline and at Week 12; Last observation carried forward (LOCF) applied to statistical analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 66 | 74 | 34 | 83 | 74
units on a scale | 2.515 (6.019) [0.75 to 3.28] | 2.405 (6.920) [0.88 to 3.27] | -0.971 (6.699) [0.7 to 3.27] | 3.530 (5.640) | 2.054 (4.800) [0.7 to 3.27]
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Only the treatment effects of 1 mg LY2452473 and 5 mg tadalafil versus 5 mg tadalafil and the treatment effects of 5 mg LY2452473 and 5 mg tadalafil versus 5 mg tadalafil were analyzed; Test type: Superiority or Other; p = 0.5, ANCOVA — The p-value was 1-sided and adjusted for multiple comparisons. The level of significance was 1-sided of 0.04; Treatment group (tx grp), baseline IIEF EF domain score, baseline testosterone level, tx grp*baseline IIEF, tx grp*testosterone level interactions
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Only the treatment effects of the treatment effects of 5 mg LY2452473 and 5 mg tadalafil versus 5 mg tadalafil and 1 mg LY2452473 and 5 mg tadalafil versus 5 mg tadalafil were analyzed; Test type: Superiority or Other; p = 0.498, ANCOVA — The p-value was 1-sided and adjusted for multiple comparisons. The level of significance was 1-sided of 0.04; The model included tx grp, baseline IIEF EF domain score, baseline testosterone level, tx grp*baseline IIEF, tx grp*testosterone level interactions

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Percentage of "Yes" Responses on the Sexual Encounter Profile (SEP) Diary
Description: The SEP diary was a participant-assessed diary with 5 questions (Q): Q1 (erection achievement), Q2 (successful penetration), Q3 (successful intercourse), Q4 (satisfied with erection), and Q5 (satisfied with sexual experience) for each sexual encounter made over a specified period of time. SEP Q1 to Q5 scores were determined as a percentage of "Yes" responses to each of the 5 questions out of all sexual attempts recorded during the time period. A higher percentage of "Yes" responses indicated better EF. Assessed was the mean change from baseline in the percentage of "Yes" responses to the SEP diary Q1 to Q5. The least squares (LS) mean was estimated from a repeated measures analysis of covariance model that included terms for treatment, visit, treatment*visit, baseline, baseline*treatment (if p-value <0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing SEP diary data at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 79 | 86 | 46 | 88 | 80
percentage of "yes" responses
  Question 1 | -0.247 (2.378) | -2.976 (2.295) | -10.711 (3.268) | 4.427 (2.168) | -1.425 (2.305)
  Question 2 | 3.175 (3.345) | 3.689 (3.227) | -7.849 (4.566) | 10.267 (3.064) | 1.844 (3.240)
  Question 3 | 9.296 (3.808) | 11.752 (3.675) | -3.800 (5.195) | 14.645 (3.489) | 2.593 (3.688)
  Question 4 | 12.935 (3.998) | 13.910 (3.854) | -1.570 (5.454) | 24.202 (3.656) | 8.857 (3.872)
  Question 5 | 13.602 (4.027) | 15.196 (3.880) | -1.956 (5.488) | 22.410 (3.683) | 9.400 (3.897)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.722, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the percentage of "Yes" responses on the SEP diary, Q1; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 1.178, Standard Error of Mean 3.312
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.634, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; LS mean of treatment difference = -1.552, Standard Error of Mean 3.253
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.147, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; LS mean of treatment difference = -4.674, Standard Error of Mean 3.218
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.020, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; LS mean of treatment difference = -7.404, Standard Error of Mean 3.157
Statistical Analysis 5: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.775, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the percentage of "Yes" responses on the SEP diary, Q2; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 1.330, Standard Error of Mean 4.658
Statistical Analysis 6: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.687, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 5]; LS mean of treatment difference = 1.844, Standard Error of Mean 4.573
Statistical Analysis 7: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.119, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 5]; LS mean of treatment difference = -7.092, Standard Error of Mean 4.535
Statistical Analysis 8: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.140, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 5]; LS mean of treatment difference = -6.578, Standard Error of Mean 4.450
Statistical Analysis 9: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.207, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the percentage of "Yes" responses on the SEP diary, Q3; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 6.703, Standard Error of Mean 5.302
Statistical Analysis 10: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.079, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 9]; LS mean of treatment difference = 9.159, Standard Error of Mean 5.206
Statistical Analysis 11: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.301, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 9]; LS mean of treatment difference = -5.349, Standard Error of Mean 5.165
Statistical Analysis 12: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.568, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 9]; LS mean of treatment difference = -2.893, Standard Error of Mean 5.067
Statistical Analysis 13: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.464, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the percentage of "Yes" responses on the SEP diary, Q4; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 4.079, Standard Error of Mean 5.566
Statistical Analysis 14: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.356, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 13]; LS mean of treatment difference = 5.054, Standard Error of Mean 5.463
Statistical Analysis 15: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.038, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 13]; LS mean of treatment difference = -11.266, Standard Error of Mean 5.418
Statistical Analysis 16: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.054, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 13]; LS mean of treatment difference = -10.292, Standard Error of Mean 5.312
Statistical Analysis 17: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.454, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the percentage of "Yes" responses on the SEP diary, Q5; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 4.202, Standard Error of Mean 5.603
Statistical Analysis 18: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.293, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 17]; LS mean of treatment difference = 5.796, Standard Error of Mean 5.499
Statistical Analysis 19: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.107, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 17]; LS mean of treatment difference = -8.808, Standard Error of Mean 5.457
Statistical Analysis 20: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.178, Mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 17]; LS mean of treatment difference = -7.214, Standard Error of Mean 5.349

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in IIEF Domain Scores (Intercourse Satisfaction, Orgasmic Function, Sexual Desire, and Overall Satisfaction)
Description: Intercourse Satisfaction (IS) domain score: sum of Questions (Q) 6, Q7, and Q8, each rated 0 (low/no satisfaction) to 5 (high satisfaction). IS domain score range: 0 to 15; lower scores denoted lower satisfaction. Orgasmic Function (OF) domain score: sum of Q9 and Q10, each rated 0 (no sexual stimulation) to 5 (almost always/always). OF domain score range: 0 to 10; lower scores denoted lower OF. Sexual Desire (SD) domain score: sum of Q11 and Q12, each rated 1 (almost never or low/no sexual desire) to 5 (almost always or very high sexual desire). SD domain score range: 2 to 10; lower scores denoted lower SD. Overall Satisfaction (OS) domain score: sum of Q13 and Q14, each rated 1 (low/no satisfaction) to 5 (high satisfaction). OS domain score range: 2 to 10; lower scores denoted lower OS. Least squares (LS) mean estimated from repeated measures analysis of variance model that included terms for treatment, visit, treatment*visit, baseline, baseline*treatment (if p-value<0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing IIEF domain scores at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 80 | 88 | 48 | 88 | 81
units on a scale
  Intercourse Satisfaction | 0.475 (0.340) | 0.514 (0.322) | -0.672 (0.463) | 1.127 (0.310) | 0.554 (0.327)
  Orgasmic Function | 0.510 (0.289) | 0.117 (0.274) | 0.160 (0.394) | 0.678 (0.264) | 0.733 (0.278)
  Sexual Desire: number analyzed (Participants) | 80 | 87 | 48 | 88 | 81
  Sexual Desire | 0.092 (0.186) | 0.001 (0.176) | -0.201 (0.253) | 0.392 (0.169) | 0.180 (0.178)
  Overall Satisfaction | 0.477 (0.247) | 0.258 (0.235) | -0.378 (0.339) | 1.206 (0.226) | 0.826 (0.238)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.867, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the IIEF IS domain score; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.079, Standard Error of Mean 0.472
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.931, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; LS mean of treatment difference = -0.039, Standard Error of Mean 0.458
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.158, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; LS mean of treatment difference = -0.652, Standard Error of Mean 0.460
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.172, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; LS mean of treatment difference = -0.612, Standard Error of Mean 0.447
Statistical Analysis 5: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.579, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the IIEF OF domain score; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.223, Standard Error of Mean 0.401
Statistical Analysis 6: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.115, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 5]; LS mean of treatment difference = -0.616, Standard Error of Mean 0.390
Statistical Analysis 7: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.668, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 5]; LS mean of treatment difference = -0.168, Standard Error of Mean 0.392
Statistical Analysis 8: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.141, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 5]; LS mean of treatment difference = -0.561, Standard Error of Mean 0.380
Statistical Analysis 9: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.734, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the IIEF SD domain score; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.088, Standard Error of Mean 0.258
Statistical Analysis 10: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.477, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 9]; LS mean of treatment difference = -0.179, Standard Error of Mean 0.251
Statistical Analysis 11: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.235, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 9]; LS mean of treatment difference = -0.300, Standard Error of Mean 0.252
Statistical Analysis 12: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.111, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 9]; LS mean of treatment difference = -0.391, Standard Error of Mean 0.245
Statistical Analysis 13: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.310, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in the IIEF OS domain score; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.349, Standard Error of Mean 0.343
Statistical Analysis 14: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.090, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 13]; LS mean of treatment difference = -0.568, Standard Error of Mean 0.334
Statistical Analysis 15: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.030, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 13]; LS mean of treatment difference = -0.729, Standard Error of Mean 0.335
Statistical Analysis 16: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.004, Mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 13]; LS mean of treatment difference = -0.948, Standard Error of Mean 0.326

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Percentage of Participants Who Return to "Normal" on the International Index of Erectile Function (IIEF) Scale (EF>25)
Description: The percentage of participants whose IIEF Erectile Function (EF) domain scores changed from ≤25 at baseline to >25 (normal) at Week 12. The IIEF EF domain score was the sum of IIEF Question (Q) 1 to Q5 and Q15. Q1 to Q5 were rated 0 (low/no EF) to 5 (high EF) and Q15 was rated 1 (no/low confidence) to 5 (high confidence). IIEF EF domain scores ranged from 1 to 30. Higher scores denoted better EF.
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population).
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 85 | 97 | 52 | 89 | 87
percentage of participants | 24.7 | 27.8 | 13.5 | 30.3 | 27.6

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in IIEF EF Domain Score Reported by Testosterone Concentration Subgroups
Description: The International Index of Erectile Function (IIEF) EF was the sum of Questions (Q) 1 to Q5 and Q15 of the IIEF Self-reported questionnaire. Q1 to Q5 were rated 0 (low/no erectile function) to 5 (high erectile function) and Q15 was rated 1 (no/low confidence) to 5 (high confidence). IIEF EF domain scores ranged from 1 to 30. Higher scores denoted better EF. Testosterone concentration subgroups were based on optimal baseline testosterone levels (<340 nanograms per deciliter [ng/dL] or ≥340 ng/dL). The least squares (LS) mean was estimated from an analysis of covariance (ANCOVA) model that included terms for treatment group, baseline, and baseline*treatment interaction (if p-value<0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing IIEF EF domain scores at baseline and at a post-baseline visit; Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 80 | 88 | 48 | 88 | 81
units on a scale
  Testosterone <340 ng/dL: number analyzed (Participants) | 43 | 54 | 28 | 54 | 47
  Testosterone <340 ng/dL | 2.523 (0.952) | 1.012 (0.848) | -1.055 (1.223) | 4.172 (0.852) | 1.935 (0.912)
  Testosterone ≥340 ng/dL: number analyzed (Participants) | 37 | 34 | 20 | 34 | 34
  Testosterone ≥340 ng/dL | 1.077 (1.019) | 3.416 (1.071) | -0.714 (1.387) | 2.217 (1.070) | 1.703 (1.063)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.656, ANCOVA — The p-value is for the change from baseline to Week 12 in the IIEF EF domain scores reported by optimal testosterone level <340 ng/dL; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.460, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.198, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.009, ANCOVA — The p-value is for the change from baseline to Week 12 in the IIEF EF domain scores reported by optimal testosterone level ≥340 ng/dL; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity
Statistical Analysis 5: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.671, ANCOVA — [p-value comment as in outcome 5, analysis 4]
Statistical Analysis 6: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.259, ANCOVA — [p-value comment as in outcome 5, analysis 4]
Statistical Analysis 7: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.441, ANCOVA — [p-value comment as in outcome 5, analysis 4]
Statistical Analysis 8: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.433, ANCOVA — [p-value comment as in outcome 5, analysis 4]

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Prostate-Specific Antigen (PSA)
Description: The least squares (LS) mean was estimated from a repeated measures analysis of covariance model that included terms for treatment, visit, treatment*visit, baseline, baseline*treatment (if p-value<0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing PSA data at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 81 | 89 | 49 | 87 | 82
nanograms per milliliter (ng/mL) | 0.162 (0.119) | -0.088 (0.109) | 0.265 (0.157) | 0.246 (0.107) | 0.032 (0.111)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.423, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 0.130
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.443, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.120
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.599, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.084
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.029, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.334

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total Cholesterol and Triglycerides
Description: as for outcome 6
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing laboratory data (total cholesterol and triglycerides) at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 81 | 90 | 49 | 88 | 82
millimoles per Liter (mmol/L)
  Total Cholesterol | -0.210 (0.076) | -0.275 (0.071) | -0.282 (0.102) | -0.086 (0.069) | -0.059 (0.072)
  Triglycerides | -0.155 (0.070) | -0.171 (0.066) | -0.067 (0.096) | -0.139 (0.063) | 0.056 (0.067)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.148, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in total cholesterol; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS Mean of treatment difference = -0.152
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.033, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; LS mean of treatment difference = -0.216
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.224, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; LS mean of treatment difference = -0.124
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.056, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; LS mean of treatment difference = -0.189
Statistical Analysis 5: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.031, Mixed model repeated measures analysis — The p-value is for the change from baseline to Week 12 in triglycerides; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.211
Statistical Analysis 6: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.017, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 5]; LS mean of treatment difference = -0.227
Statistical Analysis 7: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.866, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 5]; LS mean of treatment difference = -0.016
Statistical Analysis 8: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.726, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 5]; LS mean of treatment difference = -0.032

8. Secondary Outcome: Percent Change From Baseline to 12 Week Endpoint in High-Density Lipoprotein Cholesterol (HDL-C) and Low-Density Lipoprotein Cholesterol (LDL-C)
Description: The least squares (LS) was estimated from a repeated measures analysis of covariance model that included terms for treatment, visit, treatment*visit, baseline, baseline*treatment (if p-value<0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing laboratory data (HDL-C and LDL-C) at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 81 | 90 | 49 | 88 | 82
percent change
  HDL-C | -7.440 (1.658) | -16.974 (1.556) | -22.230 (2.243) | 1.776 (1.505) | 1.573 (1.585)
  LDL-C | -1.695 (2.479) | 0.062 (2.319) | -3.424 (3.365) | -0.066 (2.245) | -0.718 (2.367)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis — The p-value is for the percent change from baseline to Week 12 in HDL-C; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS Mean of treatment difference = -9.014
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; LS mean of treatment difference = -18.547
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; LS mean of treatment difference = -9.216
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; LS mean of treatment difference = -18.750
Statistical Analysis 5: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.776, Mixed model repeated measures analysis — The p-value is for the percent change from baseline to Week 12 in LDL-C; Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.977
Statistical Analysis 6: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.814, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 5]; LS mean of treatment difference = 0.780
Statistical Analysis 7: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.627, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 5]; LS mean of treatment difference = -1.629
Statistical Analysis 8: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.968, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 5]; LS mean of treatment difference = 0.128

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Glucose
Description: as for outcome 6
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing laboratory data (fasting glucose) at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 81 | 90 | 49 | 88 | 82
millimoles per Liter (mmol/L) | 0.153 (0.195) | -0.306 (0.183) | 0.070 (0.268) | -0.234 (0.176) | 0.158 (0.186)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.984, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS Mean of treatment difference = -0.006
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.076, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.465
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.142, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 0.387
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.776, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -0.072

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Insulin
Description: Change from baseline to 12 Week endpoint in fasting blood insulin concentration. The least squares (LS) mean was estimated from a repeated measures analysis of covariance model that included terms for treatment, visit, treatment*visit, baseline, baseline*treatment (if p-value<0.25).
Time Frame: Baseline, Week 12
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and had non-missing laboratory data (fasting insulin) at baseline and at a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: milliunits per Liter (mU/L)
Arm/Group | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 80 | 90 | 49 | 88 | 82
milliunits per Liter (mU/L) | 3.756 (2.235) | -4.501 (2.075) | -0.717 (3.068) | -3.300 (1.976) | -1.276 (2.109)
Statistical Analysis 1: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.103, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS Mean of treatment difference = 5.031
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.277, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean treatment difference = -3.225
Statistical Analysis 3: Comparison: 1 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.019, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = 7.056
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.676, Mixed model repeated measures analysis — Conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; LS mean of treatment difference = -1.201

ADVERSE EVENTS:
Groups:
- 5 mg Tadalafil, Lead-in Period: 5-mg tadalafil tablet, administered orally, once daily, during the 4-week lead-in period.
Arm/Group | 5 mg Tadalafil, Lead-in Period | 1 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 and 5 mg Tadalafil | 5 mg LY2452473 | 10 mg Tadalafil | 5 mg Tadalafil
Serious Adverse Events (participants affected / at risk) | 2/531 | 2/85 | 1/97 | 1/52 | 0/89 | 0/87
Other Adverse Events (participants affected / at risk) | 88/531 | 27/85 | 23/97 | 10/52 | 34/89 | 33/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tadalafil, Lead-in Period (N=531) | 1 mg LY2452473 and 5 mg Tadalafil (N=85) | 5 mg LY2452473 and 5 mg Tadalafil (N=97) | 5 mg LY2452473 (N=52) | 10 mg Tadalafil (N=89) | 5 mg Tadalafil (N=87)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Event resulted in death
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tadalafil, Lead-in Period (N=531) | 1 mg LY2452473 and 5 mg Tadalafil (N=85) | 5 mg LY2452473 and 5 mg Tadalafil (N=97) | 5 mg LY2452473 (N=52) | 10 mg Tadalafil (N=89) | 5 mg Tadalafil (N=87)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blood creatinine abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood testosterone abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qrs complex prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oestradiol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spider vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days